CLINICAL TRIAL: NCT02620280
Title: Neo-Adjuvant Study With the PDL1-directed Antibody in Triple Negative Locally Advanced Breast Cancer Undergoing Treatment With Nab-paclitaxel and Carboplatin
Brief Title: Neoadjuvant Therapy in TRIPle Negative Breast Cancer With antiPDL1
Acronym: NeoTRIPaPDL1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Michelangelo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FM-14-B02; 2014-005017-23 (EudraCT Number)
Record Dates: First submitted 2015-11-03; First posted 2015-12-02 (Estimated); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Invasive Ductal Breast Carcinoma
Keywords: Triple Negative Breast Cancer
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Triple Negative Breast Neoplasms | interventions — Carboplatin; Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; atezolizumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carbo-abrax, surgery, anthra (Active Comparator): Patients will receive a combination of carboplatin and abraxane as neoadjuvant treatment. Definite surgery will be performed not later than 6 weeks after the last dose of neoadjuvant therapy. Four cycles of AC or EC or FEC will then be delivered as adjuvant chemotherapy
  Interventions: Drug: Carboplatin; Drug: Abraxane; Procedure: Surgery; Drug: Anthra
- Carbo-abrax-MPDL3280A, surgery, anthra (Experimental): Patients will receive a combination of carboplatin, abraxane and MPDL3280A as neoadjuvant treatment. Definite surgery will be performed not later than 6 weeks after the last dose of neoadjuvant therapy. Four cycles of AC or EC or FEC will then be delivered as adjuvant chemotherapy
  Interventions: Drug: Carboplatin; Drug: Abraxane; Drug: MPDL3280A; Procedure: Surgery; Drug: Anthra

INTERVENTIONS:
Drug: Carboplatin — Carboplatin AUC 2 will be given i.v. on day 1 and day 8 q 3 weeks for a total of 8 cycles
  Other Names: Carboplatin Teva
Drug: Abraxane — Abraxane, 125 mg/m2 will be given i.v. on day 1 and day 8 q 3 weeks for a total of 8 cycles
  Other Names: nab-paclitaxel
Drug: MPDL3280A — MPDL3280A, 1200 mg. will be given i.v. infusion on day 1 q 3 weeks for a total of 8 cycles
  Other Names: Atezolizumab
  Arms: Carbo-abrax-MPDL3280A, surgery, anthra
Procedure: Surgery — Breast cancer surgery (breast and axilla) either conservative or radical not later than 6 weeks
Drug: Anthra — AC or EC (adriamycin or epirubicin and cyclophosphamide) or FEC (fluorouracil, epirubicin, and cyclophosphamide) on day 1 every three weeks for 4 cycles to be delivered after surgery

SUMMARY:
This study that aims to evaluate the addition of MPDL3280A (atezolizumab) to carboplatin and nab-paclitaxel in patients with early high-risk and locally advanced triple negative breast cancer. compared to the control arm of carboplatin and abraxane. Half of participants will receive MPDL3280A in combination with carboplatin and abraxane, while the other half will receive only carboplatin and abraxane.

DETAILED DESCRIPTION:
Emerging evidence shows that many breast cancers with triple negative and basal like features have infiltration by mononuclear cells and lymphocytes. Irrespective of the entity of tumor infiltration by mononuclear cells, expression of immune regulatory checkpoints such as PD-1 and its ligand B7-H1 (or PD-L1) negatively affect the results of treatments. These data suggest that a subset of patients have an ongoing immune response within the tumor micro-environment, and that PD-L1 expression is an adaptive method of tumor resistance to tumor infiltrating lymphocytes, which in turn are needed for response to chemotherapy. Overall, the data suggests a role for immune regulation of response to chemotherapy, and support the concept that blockade of immune check-points may favor the achievement of durable response by immune mechanisms themselves, and in combination with classical chemotherapy.

MPDL3280A (atezolizumab) is a human monoclonal antibody containing an engineered Fc-domain to optimize efficacy and safety that targets PD-L1 and blocks binding of its receptors, including PD-1 and B7.1. Based on these considerations, we plan to conduct a study of the combination of abraxane and carboplatin with or without PDL1-directed antibody in women with locally advanced breast cancer suitable for neoadjuvant therapy with the aim to improve event-free survival

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18 years or older with early high-risk and locally advanced or inflammatory breast cancers
2. Histologically confirmed unilateral breast cancer with invasive ductal histology not otherwise specified (NOS) of high proliferation or grade
3. HER2 negative disease
4. Negative estrogen receptor (ER) and progesterone receptor (PgR), both < 1% locally assessed
5. Representative paraffin-embedded (FFPE) tumor block taken at diagnostic biopsy for confirmation of HER2, ER and PgR eligibility, for assessment of PDL-1 expression and for further exploratory biomarker evaluation is mandatory
6. ECOG performance status 0 or 1
7. Written informed consent to participate in the trial (approved by the Institutional Review Board [IRB]/ Independent Ethics Committee [IEC]) obtained prior to any study specific screening procedures
8. Willing and able to comply with the protocol
9. Consent to the collection of blood samples
10. For women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to remain abstinent or use single or combined contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 90 days after the last dose of study drug.

Exclusion Criteria:

1. Evidence of bilateral breast cancer or metastatic disease (M1)
2. Cases with an histology different from invasive ductal NOS of high proliferation or grade
3. Patients with HER2-positive disease according to ASCO/CAP guidelines 2013
4. Pregnant or lactating women. Documentation of a negative pregnancy test must be available for premenopausal women with intact reproductive organs and for women less than one year after the last menstrual cycle
5. Previous treatment with chemotherapy, hormonal therapy or an investigational drug for any type of malignancy
6. Previous investigational treatment for any condition within 4 weeks of randomization date
7. Administration of a live, attenuated vaccine within 4 weeks before cycle 1 Day 1 or anticipation that such a live attenuated vaccine will be required during the study
8. Previous or concomitant invasive malignancy of any other type or previous invasive breast cancer. Patients with curatively treated basal cell carcinoma of the skin or in situ cervix cancer are generally eligible
9. Pre-existing motor or sensory neuropathy of grade > 1 for any reason
10. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
11. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the MPDL3280A formulation
12. Patients with prior allogeneic stem cell or solid organ transplantation
13. History of autoimmune disease including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Bell's palsy, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis
14. History of idiopathic pulmonary fibrosis (including bronchiolitis obliterans with organizing pneumonia) or evidence of active pneumonitis on screening chest computed tomography scan
15. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, fatty liver, and inherited liver disease
16. History of HIV infection, active hepatitis B (chronic or acute), or hepatitis C infection. Patients with past or resolved hepatitis B infection (defined as having a negative HBsAg test and a positive hepatitis B core antigen [anti-HBc] test) are eligible.

Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction assay (PCR) is negative for HCV RNA 17. Active tuberculosis 18. Severe infections within 4 weeks prior to cycle 1 Day 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia. Signs or symptoms of significant infection within 2 weeks prior to cycle 1 Day 1 19. Received oral or IV antibiotics within 2 weeks prior to Cycle 1 Day 1 20. Other serious illness or medical condition including: history of documented congestive cardiac failure; New York Heart Association (NYHA) Class II or greater CHF; angina pectoris requiring anti-anginal medication or unstable angina within 6 months prior to cycle 1 Day 1; evidence of transmural infarction on ECG; myocardial infarction stroke or transient ischemic attack (TIA) within 6 months prior to cycle 1 Day 1; poorly controlled hypertension (e.g. systolic >180 mm Hg or diastolic >100 mm Hg; however, patients with hypertension which is well controlled on medication are eligible); clinically significant valvular heart disease; high-risk uncontrolled arrhythmias 21. Patients with a history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and precluding informed consent or adversely affecting compliance with study drugs 22. Serious uncontrolled infections (bacterial or viral) or poorly controlled diabetes mellitus 23. Abnormal baseline hematological values 24. Abnormal baseline laboratory tests for serum total bilirubin, liver function tests, alkaline phosphatase, serum creatinine, INR and aPTT 25. Baseline left ventricular ejection fraction (LVEF) < 50% by echocardiography or multi-gated scintigraphic scan (MUGA) 26. Major surgical procedure within 28 days prior to cycle 1 Day 1 or anticipation of need for a major surgical procedure during the course of the study 27. Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist®) within 4 weeks prior to cycle 1 Day 1 or at any time during the study.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2016-04; Primary Completion 2024-01 (Actual); Study Completion 2024-01-07 (Actual)

PRIMARY OUTCOMES:
Event Free Survival (EFS) | 5 years after the randomization of the last patient
  To compare EFS (disease progression while on neoadjuvant therapy or disease recurrence after surgery) in the two study arms

SECONDARY OUTCOMES:
Pathological complete response (pCR) | At surgery, an expected average of 34 weeks after the randomization of the last patient
  Assess the rate of pCR defined as ypT0-ypTis ypN0 at surgery in the two treatment arms
Clinical objective response | Participants will be followed for the duration of neoadjuvant therapy, an expected average of 26 weeks
  Assess the clinical response rate after neoadjuvant therapy
Distant Event Free Survival (DEFS) | 5 years after the randomization of the last patients
  To compare the DEFS, defined as the occurrence of distant disease progression while on neoadjuvant therapy or distant recurrence after surgery in the two treatment arms
Number of participants with adverse events as a Measure of Safety and Tolerability | Participants wil be followed for up to 5 years from the last randomized patient
  Number of participants with Adverse Events and related grade

CONTACTS AND LOCATIONS:
Overall Officials: Luca Gianni, MD, Study Chair — Ospedale San Raffaele
Locations (41):
- Austria (2):
  - Brustgesundheitzentrum Tirol, Univ. Frauenklinik Innsbruck, Innsbruck
  - Universitätsklinik für Innere Medizin III, mit Hämatologie, internistischer Onkologie, Hämostaseologie, Infektiologie, Rheumatologie und Onkologisches Zentrum, Salzburg
- Germany (10):
  - Klinikum Augsburg International Patient Service, Augsburg
  - Frauenarzt-Zentrum-Zehlendorf, Berlin
  - Augusta-Kranken-Anstalt gGmbH Klinik für Hämatologie, Onkologie & Palliativmedizin, Bochum
  - Uniklinik Köln Klinik und Poliklinic für Frauenheilkunde und Geburtshilfe Brestzentrum, Cologne
  - Brustzentrum St. Elisabeth-Krankenhaus, Cologne
  - Bethanien-Krankenhaus Onkologisches Zentrum, Frankfurt
  - Markus Krankenhaus Klinik für Gynäkologie und Geburtshilfe, Frankfurt
  - Gynäkologisch-Onkologische Praxis, Hanover
  - NCT Nationales Centrum für Tumorerkrankungen, Heidelberg
  - Interdisciplinary Oncology Center (IOZ), München
- Ireland (5):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
  - University Hospital Waterford, Waterford
- Italy (10):
  - Policlinico S. Orsola Malpoghi, Bologna
  - Istituto per la Ricerca sul Cancro, Candiolo
  - IST San Martino, Genova
  - Istituto Toscano Tumori Ospedale Misericordia, Grosseto
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia, Milan
  - Ospedale Luigi Sacco, Milan
  - Arcispedale Santa Maria Nuova - A.O. Reggio Emilia, Reggio Emilia
  - Ospedale Santa Maria della Misericordia, Udine
- Russia (3):
  - Russian Cancer Research Center named after N.N.Blokhin, Moscow
  - Petrov Research Institute of Oncology, Department of Breast Cancer, Saint Petersburg
  - Road clinical hospital of OJSC "Russian Railways, Saint Petersburg
- Spain (6):
  - Hospital Duran i Reynal Institut Català d'Oncologia, L'Hospitalet de Llobregat
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de octubre, Madrid
  - Hospital Universitario HM Sanchinarro, Centro Integral Oncologico Clara Campal (CIOCC), Madrid
  - Hospital Clinico Universitario de Valencia Servicio de Onco-Hematologia, Valencia
  - Hospital Miguel Servet, Zaragoza
- Taiwan (5):
  - C. Christian Hospital Taiwan, Changhua
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - China Medical University Hospital No.2, Taichung
  - National Taiwan University Hospital, Taipei
  - Veteran General Hospital Taipei, Taipei

REFERENCES:
- [Derived] Gianni L, Huang CS, Egle D, Bermejo B, Zamagni C, Thill M, Anton A, Zambelli S, Bianchini G, Russo S, Ciruelos EM, Greil R, Semiglazov V, Colleoni M, Kelly C, Mariani G, Del Mastro L, Maffeis I, Valagussa P, Viale G. Pathologic complete response (pCR) to neoadjuvant treatment with or without atezolizumab in triple-negative, early high-risk and locally advanced breast cancer: NeoTRIP Michelangelo randomized study. Ann Oncol. 2022 May;33(5):534-543. doi: 10.1016/j.annonc.2022.02.004. Epub 2022 Feb 17. PMID 35182721
- [Derived] Perez-Garcia J, Soberino J, Racca F, Gion M, Stradella A, Cortes J. Atezolizumab in the treatment of metastatic triple-negative breast cancer. Expert Opin Biol Ther. 2020 Sep;20(9):981-989. doi: 10.1080/14712598.2020.1769063. Epub 2020 May 25. PMID 32450725